CLINICAL TRIAL: NCT01068639
Title: IMprove PAtient Compliance sTudy: An Observational, Cross-sectional Study on Children Treated With Growth Hormone in France
Brief Title: An Observational Study on Treatment Compliance by Children Treated With Growth Hormone
Acronym: IMPACT
Status: Withdrawn | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3787; U1111-1113-2490 (Other: WHO)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Behavioral: No treatment given

INTERVENTIONS:
Behavioral: No treatment given — No treatment given to study participants, only behaviorial patterns with respect to treatment compliance is observed.

SUMMARY:
This study is conducted in Europe. This observational study aims at evaluating compliance with growth hormone treatment in children and identifying factors influencing compliance.

ELIGIBILITY:
Inclusion Criteria:

* Child treated for at least one year with growth hormone any growth hormone product
* Followed by the participating paediatrician for at least 1 year.

Exclusion Criteria:

* Refusal to participate
* Child and/or parent unable to give consent or fill out the questionnaires
* Child participating in a therapeutic trial

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children treated for at least one year with growth hormone with any growth hormone product whatever the reason for prescription
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Average number of injections omitted during the previous month | measured over the past 2 months (retrospective data collection)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com